CLINICAL TRIAL: NCT04114071
Title: TOSS Feasibility + Fitbit Community = Reduced Obesity in Older Black Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Pamela G Bowen PhD, CRNP, FNP-BC, BBA, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB 300004159; U54MD000502 (NIH)
Record Dates: First submitted 2019-10-01; First posted 2019-10-03 (Actual); Results first posted 2022-10-14 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Obesity
Keywords: physical activity; older Black women; overweight; obesity; text messages
MeSH Terms: conditions — Obesity; Motor Activity; Overweight

STUDY DESIGN:
Intervention Model Description: The researchers hypothesize that older overweight or obese Black women who participate in the PA intervention group (TOSS text messages plus Fitbit) will show increases in self-report and objective (assessed by accelerometer and a Fitbit) PA behaviors compared to the control group.
Who Masked: Participant
Masking Description: All participants will receive text messages during the 12-week intervention but the frequency, the content of the messages will be different for the control and intervention groups, and these differences will not be discussed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Activity intervention group (Experimental): Older overweight or obese Black women who participate in the physical activity intervention group will receive a daily text message from the TOSS study for 12 weeks, a Fitbit device plus have access to the Fitbit community option on their Fitbit app as an opportunity for virtual peer support. They will also receive an instruction pamphlet that describes the health benefits of regular physical activity (PA), safety instructions for PA, the national PA guidelines for older adults, suggested strategies to increase number of steps and an accelerometer pre and post-intervention.
  Interventions: Behavioral: TOSS Feasibility + Fitbit Community = Reduced Obesity in Older Black Women
- Control group (Active Comparator): The control will only receive a weekly neutral text message during the 12-week intervention. For this project, a neutral text message is defined as a message that only provides facts about a topic.They will also receive a Fitbit device, an instruction pamphlet that describes the health benefits of regular physical activity (PA), safety instructions for PA, the national PA guidelines for older adults, suggested strategies to increase number of steps and an accelerometer pre and post-intervention
  Interventions: Behavioral: TOSS Feasibility + Fitbit Community = Reduced Obesity in Older Black Women

INTERVENTIONS:
Behavioral: TOSS Feasibility + Fitbit Community = Reduced Obesity in Older Black Women — See arm description

SUMMARY:
The primary goal of this proposed physical activity (PA) intervention is to develop a realistic and an economical intervention to promote regular PA among older, overweight or obese Black women. Physical inactivity is prevalent among older Black women and this lifestyle behavior is both a destructive and expensive public health issue. Because many in this population do not engage in sufficient amounts of regular PA, this group miss the cardio-protective effects that may reduce many chronic conditions that disproportionately affect Blacks such as hypertension, diabetes, and obesity. The proposed obesity-reduction intervention is aligned with Stage 1 of the National Institute on Aging Stage Model for Behaviors Interventions Development. For the proposed hypothesis, the investigators propose a 2-group randomized controlled pilot, feasibility study in which 30 women will be randomized to receive either the TOSS PA Text messages Plus Fitbit community or the Control group and followed for 12 weeks to detect intervention effect.

ELIGIBILITY:
Inclusion Criteria:

* Black women
* 60 years and older
* Have a BMI ≥ 25 kg/m2
* Do not meet the weekly 150 minutes of physical activity (PA)
* No health conditions that would prevent or limit PA or walking
* Able to read text messages
* Access to a mobile phone with text receiving capability
* Mobile phone with ability to download a Fitbit app.

Exclusion Criteria:

* Currently participating in another PA promotion program
* Non-English speaking
* A contraindication to exercise as indicated by the PA Readiness Questionnaire (PAR-Q) unless written permission was provided from the participant's primary care provider.

Min Age: 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-07-16 (Actual); Primary Completion 2020-12-28 (Actual); Study Completion 2020-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela G. Bowen, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Pamela G. Bowen, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bowen PG, Affuso O, Opoku-Agyeman W, Mixon VR, Clay OJ. Texting Older Sisters to Step to Manage Obesity in Older Black Women: A Feasibility Study. Am J Prev Med. 2022 Jul;63(1 Suppl 1):S56-S66. doi: 10.1016/j.amepre.2022.03.014. PMID 35725141

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Physical Activity Intervention Group | Control Group
Started | 15 | 15
Completed | 14 | 15
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Physical Activity Intervention Group | Control Group | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 6 | 13
  >=65 years | 8 | 9 | 17
Age, Continuous [Mean (Full Range); unit: years] | 64.67 [60 to 70] | 65.33 [60 to 70] | 65 [60 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 15 | 30
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 15 | 30
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 34.52 (4.20) | 35.33 (5.95) | 34.93 (5.08)
hemoglobin A1c [Mean (Standard Deviation); unit: percent of gylcosylated hemoglobin] | 6.18 (2.18) | 6.39 (0.58) | 6.29 (1.57)
weight [Mean (Standard Deviation); unit: lbs] | 209.7 (32.76) | 212.3 (41.22) | 211.02 (36.61)
Steps per day [Mean (Standard Deviation); unit: Daily steps] | 6207.85 (4315.71) | 6506.85 (3480.18) | 6357.35 (3855.08)

OUTCOME MEASURES:

1. Primary Outcome: Change in Physical Activity Behaviors From Baseline to 12 Weeks
Description: number of steps
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: change in daily steps (baseline - post)
Arm/Group | Physical Activity Intervention Group | Control Group
Number analyzed (Participants) | 15 | 15
change in daily steps (baseline - post) | -736.71 (4315.71) | 218.79 (3480.18)
Statistical Analysis 1: Comparison: Physical Activity Intervention Group vs Control Group; Test type: Equivalence — An independent sample t tests was used to examine the difference score for each of the four outcome measures of interest (steps, WC, weight, and HbA1c) between intervention and control groups; p < 0.05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 12 weeks
Groups:
- Physical Activity Intervention Group: Older overweight or obese Black women who participate in the physical activity intervention group will receive a daily text message from the TOSS study for 12 weeks, a Fitbit device plus have access to the Fitbit community option on their Fitbit app as an opportunity for virtual peer support. They will also receive an instruction pamphlet that describes the health benefits of regular physical activity (PA), safety instructions for PA, the national PA guidelines for older adults, suggested strategies to increase number of steps and an accelerometer pre and post-intervention.
  TOSS Feasibility + Fitbit Community = Reduced Obesity in Older Black Women: See arm description
  No adverse events in this group.
- Control Group: The control will only receive a weekly neutral text message during the 12-week intervention. For this project, a neutral text message is defined as a message that only provides facts about a topic.They will also receive a Fitbit device, an instruction pamphlet that describes the health benefits of regular physical activity (PA), safety instructions for PA, the national PA guidelines for older adults, suggested strategies to increase number of steps and an accelerometer pre and post-intervention
  TOSS Feasibility + Fitbit Community = Reduced Obesity in Older Black Women: See arm description
  No adverse events in this group.
Arm/Group | Physical Activity Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-11-12): https://cdn.clinicaltrials.gov/large-docs/71/NCT04114071/Prot_000.pdf
  • Informed Consent Form (2019-11-12): https://cdn.clinicaltrials.gov/large-docs/71/NCT04114071/ICF_001.pdf